CLINICAL TRIAL: NCT04290442
Title: A Prospective Randomized Parallel Study to Compare Post-operative Pain Control With Addition of Sensory Posterior Articular Nerve Block to Adductor Canal Block (SPANK) and Intraoperative Periarticular Infiltration in Total Knee Arthroplasty.
Brief Title: Adductor Canal Vs Adductor Canal Plus SPANK Block for Postoperative Pain in Knee Arthroplasty Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: initially cessation due to covid, then fellow doing the study graduated with no time to complete the study; will take up again if a current fellow takes on the project
Sponsor: Bruce Ben-David (Other)
Responsible Party: Sponsor-Investigator, Bruce Ben-David, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19120105
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Arthroplasty, Replacement, Knee; Anesthesia, Conduction; Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The study will be conducted as prospective, randomized, single blinded, parallel trial at the University of Pittsburgh Medical Center (UPMC) Shadyside Hospital.
Who Masked: Outcomes Assessor
Masking Description: At the office of acute pain management, one member of the research team will be responsible for providing the anesthesiologist in charge of performing the block with a sealed envelope. Each envelope will be labeled with a number corresponding to a matching number labeled on each patient binder. This envelope will contain the information regarding the block type based on randomization to be administered to the patient. Once the anesthesiologist knows which block he is going to administer, he will reseal the envelope and return it to the research team member. This process will allow only the anesthesiologist performing the block to have knowledge of the block type he or she is administering, keeping research team members blinded. The envelopes and binders will be kept by the principal investigator in a safe place and only reopened to be analyzed at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adductor canal block (ACB) (Active Comparator)
  Interventions: Procedure: adductor canal block; Drug: Ropivacaine
- Adductor canal block plus SPANK block (Experimental)
  Interventions: Procedure: adductor canal block; Procedure: SPANK; Drug: Ropivacaine

INTERVENTIONS:
Procedure: adductor canal block — The block is performed in supine position under ultrasound guidance using 22 G Touhy needle advanced in plane and 15 cc of 0.5% Ropivacaine ( local anesthetic) with dexmedetomidine 20-30 mcg depending on the age of the patient is injected at midthigh level lateral to the femoral artery in adductor canal to provide sensory blockade to the anterior aspect of the knee.
Procedure: SPANK — SPANK: The block is performed in supine position, using 22 G Touhy needle, under ultrasound guidance, needle is advanced in plane to posteromedial shaft of femur taking care to avoid popliteal artery, and 0.5% ropivacaine 15 cc, dexmedetomidine 20-30mcg and dexamethasone 4 mg is injected into inner thigh above the knee provide sensory block to posterior aspect of the knee.
  Arms: Adductor canal block plus SPANK block
Drug: Ropivacaine — ropivacaine 0.5% will be use in the block

SUMMARY:
This study will prospectively investigate the efficacy of Adductor canal block with periarticular infiltration Vs Adductor canal block, Periarticluar infiltration and Sensory posterior articular nerve of the knee block in patients undergoing total knee arthroplasty. The study will aid in answering question whether SPANK block is an effective adjunct in preventing posterior knee pain without causing motor blockade.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA)is a common orthopedic surgical procedure. Optimal pain control is necessary for early recovery and discharge. TKA is considered one of the more painful surgical procedures, peripheral nerve blocks and multimodal analgesia are incorporated into clinical practice to provide patient comfort, decrease postoperative opioid requirement, facilitate early ambulation and enhance patient satisfaction.Adductor canal nerve block (ACB) and intraoperative periarticular infiltration (PAI) are routine clinical practice followed at our institute for postoperative pain control. Although ACB provided analgesia to peripatellar and anterior intra-articular aspect of knee joint, it does not relieve posterior knee pain which can be moderate to severe in intensity. Many techniques have been employed for posterior knee pain including sciatic nerve block and infiltration between popliteal artery and posterior capsule of the knee joint (IPACK) with limited success. Sciatic nerve block is considered gold standard but is rarely used due to associated motor weakness, which may delay ambulation and decrease participation in physical therapy postoperatively . In recent times IPACK block has gained popularity but there are concerns about local anesthetic injection close to surgical field and total dose of local anesthetic exceeding the recommended amount if combined with periarticular infiltration as is the practice at our institute.

SPANK block was described in 2015 by Kardash et al for posterior knee pain while sparing motor function. The block is performed at the level of femoral shaft above the femoral epicondyle, on the medial side of the leg, with needle positioned just superficial to posteromedial femoral periosteum and 15 ml of local anesthetic is injected, decreasing concerns for local anesthetic toxicity, and invasiveness close to surgical field as compared to IPACK block which requires 30 ml of local anesthetic.

Efficacy of SPANK block has been demonstrated as rescue analgesic for posterior knee pain after TKA, and a trial is underway to evaluate efficacy of ACB an SPANK block versus ACB alone [5].There is no literature evaluating benefit of SPANK block when added to ACB and PAI which is a standard practice.

If SPANK block proves to be effective in controlling posterior knee pain, with motor sparing effect it can help reduce postoperative opioid requirement, help achieve same day discharge and prove to be another small step towards fighting opioid epidemic.

Hence, we propose this study to evaluate added benefit of SPANK block to ACB and PAI with regards to postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 19 and 90 years old. BMI 18-45 ASA class I-II-III

Exclusion Criteria:

Simultaneous bilateral TKA.

History of substance abuse.

BMI >45.

Patients that did not received Intrathecal anesthesia.

Infection at the site of injection (either for spinal or PNB).

Pregnancy.

Non english speaking or inability to participate in the study.

Patients with coagulopathy or With INR >1,5 the day of the surgery.

Pharmacologic coagulopathy: patients on xarelto, plavix, or any kind of "Blood Thinners".

Chronic steroid use: patients with consumption of steroid for more than 3 months.

Chronic pain: pain for more than 3 months.

Chronic opiate use : consumption of opioids for more than 3 months.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain score using Numerical rating Scale (NRS) with ambulation at 24 hours after total knee arthroplasty | At 24 hours after surgery
  Patient will describe the pain experienced after surgery on a scale from 1-10 being 10 the worst pain ever experienced, this will be registered in the format designed for this purpose and at the end of the study will be analyzed

SECONDARY OUTCOMES:
Pain scores at rest and with movement at 6, 12 and 24 hours after the surgery measured using Numerical Rating Scale (NRS). | It will be measured at 6 hours, 12 hours, 24 hours after surgery
  Patient will describe the pain experienced after surgery in rest and in movement at 6,12,24 hours on a scale from 1-10 being 10 the worst pain ever experienced.
Time to first opioid Consumption | During the first 24 after surgery
  The amount of time measured from the end of the surgery when the patient leaves the operating room to the time when they receive their first dose of any opioid medication.
Opioid consumption | During the first 24 after surgery
  will be measured using morphine equivalents during first 24 hours after knee surgery, starting when the patient leaves the operating room
Extent of motor blockade in various lower extremity muscle groups | During the first 24 after surgery
  This outcome will be reported by physical therapy on medical records
Time that the patient takes to walk 100 feet after surgery | During the first 24 after surgery
  This outcome will be reported by physical therapy on medical records
Patient satisfaction with the pain management strategy provided after first 24 hours. | During the first 24 after surgery
  patient satisfaction survey will be answered by the patient at 24 hours after surgery. This questionnaire will have a score of satisfaction from1-5, being 5 the maximum satisfaction experienced by the patient.
Local anesthetic toxicity reported in the medical records if is present. | During the first 24 after surgery
  Local Anesthetic Toxicity is defined by symptoms such as metallic taste, tinnitus, drowsiness, after administering a dose of local anesthetics.This will be reported in the medical record and by the physician on call.t We will measure the number of participants that present these kind of symptoms if any.
Nausea and vomiting | During the first 24 after surgery
  The presence or absence of nausea and vomiting, and the number of episodes during the first 24 hours after surgery.The outcome assessor will ask directly to the patient about this symptoms.we will measure the number of patients that report these symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ben-David, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Karlsen AP, Wetterslev M, Hansen SE, Hansen MS, Mathiesen O, Dahl JB. Postoperative pain treatment after total knee arthroplasty: A systematic review. PLoS One. 2017 Mar 8;12(3):e0173107. doi: 10.1371/journal.pone.0173107. eCollection 2017. PMID 28273133
- [Background] Vora MU, Nicholas TA, Kassel CA, Grant SA. Adductor canal block for knee surgical procedures: review article. J Clin Anesth. 2016 Dec;35:295-303. doi: 10.1016/j.jclinane.2016.08.021. Epub 2016 Oct 11. PMID 27871547
- [Background] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648